CLINICAL TRIAL: NCT01938729
Title: Phase I Study of Hepatic Arterial Infusion With Floxuridine and Dexamethasone in Combination With Gemcitabine as Adjuvant Treatment After Resection of Intrahepatic Cholangiocarcinoma
Brief Title: Hepatic Arterial Infusion With Floxuridine and Dexamethasone in Combination With Gemcitabine as Adjuvant Treatment After Resection of Intrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ohio State University (Other); University of Texas Southwestern Medical Center (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-148
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Intrahepatic Cholangiocarcinoma; Peripheral Cholangiocarcinoma; Cholangiolar Carcinoma; Cholangiocellular Carcinoma) (ICC)
Keywords: HEPATIC ARTERIAL INFUSION; FLOXURIDINE; DEXAMETHASONE; GEMCITABINE; Pump; 13-148
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Hepatectomy; Floxuridine; Dexamethasone; Gemcitabine

ARMS (1):
- HAI with FLOXURIDINE & DEXAMETHASONE & GEMCITABINE (Experimental): This is an open-label single arm study. multi-institution phase I dose escalating trial of adjuvant HAIP FUDR and Gemcitabine chemotherapy after curative resection of ICC. Hepatectomy with or without bile duct reconstruction and pump placement are performed. The patients will start therapy 4 weeks postoperatively. They will receive HAI FUDR/Dex and systemic gemcitabine in the following dose escalation levels of gemcitabine. The dose of HAI FUDR will be fixed. A classic 3+3 cohort dose escalation scheme will be used to identify the MTD of the combination.
  Level 1: Systemic gemcitabine 650mg/m^2 Day 1 and 15 and HAI FUDR/Dex 0.12mg/kg/day Day 1-14 Level 2.Systemic gemcitabine 800mg/m^2 Day 1 and 15 HAI FUDR/Dex 0.12 mg/kg/day Day 1-14 Level 3. Systemic gemcitabine 1000mg/m^2 Day 1 and 15 HAI FUDR/Dex 0.12 mg/kg/day Day 1-14
  Interventions: Procedure: Liver resection and placement of hepatic artery infusion pump; Drug: FLOXURIDINE; Drug: DEXAMETHASONE; Drug: GEMCITABINE

INTERVENTIONS:
Procedure: Liver resection and placement of hepatic artery infusion pump
Drug: FLOXURIDINE
Drug: DEXAMETHASONE
Drug: GEMCITABINE

SUMMARY:
This is a Phase I study, which means we want to find out what effects, good and/or bad, this combination of drugs may have on the patient and the liver cancer at different dose levels. All patients will have an operation to remove tumors in the liver and may have a pump placed in their abdomen.

On this study, both drugs given have been used in other patients for treatment of cholangiocarcinoma and other gastrointestinal cancers. Both drugs are approved by the food and drug administration (FDA) for treatment of liver cancer, but the two drugs have only been combined in a few patients.

That means that in this trial we also want to find out if this combination is safe.

The study will also evaluate if this treatment works in delaying or stopping the cancer from coming back after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intrahepatic cholangiocarcinoma (also variously reported as peripheral cholangiocarcinoma, cholangiolar carcinoma or cholangiocellular carcinoma) (ICC). Confirmation of the diagnosis must be made at MSKCC or at the participating institution prior to initiating protocol therapy.
* Technically resectable, single tumors of any size, tumors with satellite nodules within 2 cm of the primary tumor that are resectable. Limited and resectable multi-focal disease (less than 4 tumors technically resectable).
* Patients with elevated liver function tests including jaundiced patients (due to tumor) can be selectively operated on without resolution of jaundice preoperatively according to the judgment of the operating surgeon
* Patients must have a KPS > 80% and be considered candidates for general anesthesia, hepatic resection and hepatic artery pump placement.
* Laboratory values within 14 days before registration must be:
* Serum albumin must be >2.5 g/dl
* Creatinine must be < 1.8 mg/dL
* WBC must be >3500 cells/mm3
* Platelet count must be >100,000/mm3
* International normalized ratio (INR) must be less than 1.5 in patients not on Coumadin therapy
* Technically resectable, single tumors of any size, tumors with satellite nodules within 2 cm of the primary tumor that are resectable. Limited and resectable multi- focal disease (less than 4 tumors technically resectable).
* Patients with elevated liver function tests including jaundiced patients (due to tumor) can be selectively operated on without resolution of jaundice preoperatively according to the judgment of the operating surgeon
* Age >18 years
* Patients must be able to understand and sign informed consent
* Prior chemotherapy is allowed

Exclusion Criteria:

* Prior treatment with HAI chemotherapy
* Extrahepatic metastases including nodal disease
* Prior external beam radiation therapy to the liver
* Diagnosis of sclerosing cholangitis
* Diagnosis of Gilbert's disease
* Clinical ascites
* Hepatic encephalopathy
* Patients who have radiographic evidence of esophageal varices or history of variceal hemorrhage
* Patients with occlusion of the main portal vein or of the right and left portal branches
* Patients that have concurrent malignancies (except localized basal cell or squamous cell skin cancers)
* Female patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Safety and Toxicity | 1 year
  All toxicities will be rated as per the NCI Common Toxicity Criteria (CTC AE version 4.0) except neurosensory and hepatic enzyme toxicities related to intrahepatic pump therapy.

SECONDARY OUTCOMES:
Recurrence Free Survival | 1 year
  we will evaluate the recurrence-free survival of patients in this trial using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center Sleepy Hollow, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/